CLINICAL TRIAL: NCT00835133
Title: Biospecimen Resource for Familial Pancreas Research, a Data and Tissue Registry (Also Known as a Bio-repository, Bio-bank, Data and Tissue Database, Data and Tissue Bank, Etc.) to Help Advance Research in Familial Pancreas Disease
Brief Title: Collecting Blood and Tissue Samples From Family Members of Patients With Pancreatic Diseases, Pancreatic Cancer, and Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shounak Majumder, Principal Investigator, Mayo Clinic
Other Study IDs: 355-06; R01CA097075-08 (NIH); CDR0000613097 (Registry Identifier: NCI)
Record Dates: First submitted 2009-01-31; First posted 2009-02-03 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Familial Pancreatic Cancer
Keywords: family; history; pancreas; cancer; melanoma; genetic
MeSH Terms: conditions — Pancreatic carcinoma, familial; Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 10mL plasma tubes and two 10mL serum tubes collected. DNA extracted from blood lymphocytes.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: biologic sample preservation procedure — one blood sample
Other: medical chart review — confirmation of cancer diagnosis
Other: survey administration — at baseline enrollment and 12 months post-enrollment

SUMMARY:
RATIONALE: Collecting and storing samples of blood and tissue from family members of patients with cancer to test in the laboratory may help the study of cancer in the future.

PURPOSE: This clinical trial is collecting blood and tissue samples from family members of patients with pancreatic disease, pancreatic cancer, and melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect clinical history, family history, and blood and/or tissue samples from family members of patients diagnosed with pancreatic diseases, pancreatic cancer, or melanoma.
* To learn whether inherited factors increase the risk of pancreatic diseases, pancreatic cancer, or other cancers.

OUTLINE: Study participants undergo collection of blood and/or tissue samples as well as survey data for inclusion in a familial data and tissue registry. Participants complete two baseline surveys regarding their personal, family, health, and environmental exposure histories and regarding their opinions on cancer and cancer screening. Patients also complete a follow-up survey at 1 year and undergo review of their medical records.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Has at least 2 blood relatives with pancreatic cancer (both must be related)
  * Has at least 1 blood relative with pancreatic cancer and 1 with melanoma (both must be related)

PATIENT CHARACTERISTICS:

* Mentally competent and able to provide informed consent
* Able to understand and read English

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Familial pancreatic cancer kindred
Sampling Method: Non-Probability Sample
Enrollment: 1122 (Actual)
Dates: Start 2002-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Collection of familial data and biospecimens in a data and tissue repository for familial pancreas research | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Shounak Majumder, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials